CLINICAL TRIAL: NCT06789913
Title: A Phase 2 Study of Mutant-selective PI3Kα Inhibitor, RLY-2608, in Adults and Children With PIK3CA Related Overgrowth Spectrum and Malformations Driven by PIK3CA Mutation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Relay Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RLY-2608-201; 2024-518895-30-00 (EU CTIS Number)
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: PIK3CA-Related Overgrowth Spectrum (PROS); Lymphatic Malformations; Vascular Malformations; PIK3CA Mutation; CLOVES Syndrome; Klippel Trenaunay Syndrome; Megalencephaly-capillary Malformation Polymicrogyria Syndrome (MCAP)
MeSH Terms: conditions — Lymphatic Abnormalities; Vascular Malformations; Congenital Lipomatous Overgrowth, Vascular Malformations, and Epidermal Nevi; Klippel-Trenaunay-Weber Syndrome; Megalencephaly cutis marmorata telangiectatica congenita

STUDY DESIGN:
Intervention Model Description: Part 1: Dose selection: Participants ≥12 years old with PROS or malformations with PIK3CA mutation (Group 1) will be randomly assigned to a selected dose of RLY-2608 in an open-label fashion, stratified based on prior treatment with alpelisib. Groups 2 (6 to <12 years old) and 3 (2 to <6 years old): RLY-2608 will be studied in pediatric participants in a dose escalation design.
  Part 2: Part 2 will explore the clinical activity of RLY-2608 at 1 or more adult, adolescent, and pediatric recommended Phase 2 dose (RP2D) in various populations of participants with PROS and malformations associated with PIK3CA mutations in an open-label basket trial design.
  Part 3: In Part 3, adult (>18 yo), and adolescent and pediatric (6 to <18 yo) participants with PROS and malformations with PIK3CA mutation will be randomized to receive RLY-2608 at the Group 1 and 2 RP2Ds versus placebo. Randomization will be stratified based on indication, and prior systemic therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part 1, Group 1 (Experimental): RLY-2608 for patients ≥12 years old with PROS or malformations with PIK3CA mutation. Multiple doses of RLY-2608 for oral administration.
  Interventions: Drug: RLY-2608
- Part 1, Group 2 (Experimental): RLY-2608 for participants 6 to <12 years old with PROS or malformations with PIK3CA mutation.
  RLY-2608 will be studied in pediatric participants in a dose escalation design.
  Interventions: Drug: RLY-2608
- Part 1, Group 3 (Experimental): Part 1, Group 3: RLY-2608 for participants 2 to <6 years old with PROS or malformations with PIK3CA mutation.
  RLY-2608 will be studied in pediatric participants in a dose escalation design.
  Interventions: Drug: RLY-2608
- Part 2, Group 1 (Experimental): Dose expansion single-arm cohorts for various subpopulations of participants ≥12 years old with PROS or malformations with PIK3CA mutation.
  Oral dose of RLY-2608 as determined during Part 1.
  Interventions: Drug: RLY-2608
- Part 2, Group 2 (Experimental): Dose expansion cohorts for participants 6 to <12 years old with PROS or malformations with PIK3CA mutation.
  Oral dose of RLY-2608 as determined during Part 1.
  Interventions: Drug: RLY-2608
- Part 2, Group 3 (Experimental): Dose expansion cohorts for participants 2 to <6 years old with PROS or malformations with PIK3CA mutation.
  Oral dose of RLY-2608 as determined during Part 1.
  Interventions: Drug: RLY-2608
- Part 3, Arm 1 (Experimental): Adult (>18 yo), and adolescent and pediatric (6 to <18 yo) participants with PROS and malformations with PIK3CA mutation will be randomized to receive RLY-2608 at oral dose determined during Part 1/2 versus placebo.
  Interventions: Drug: RLY-2608
- Part 3, Arm 2 (Placebo Comparator): Adult (>18 yo), and adolescent and pediatric (6 to <18 yo) participants with PROS and malformations with PIK3CA mutation will be randomized to receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RLY-2608 — RLY-2608 is a mutant-selective, oral PI3Kα inhibitor.
  Arms: Part 1, Group 1; Part 1, Group 2; Part 1, Group 3; Part 2, Group 1; Part 2, Group 2; Part 2, Group 3; Part 3, Arm 1
Drug: Placebo — RLY-2608 matched-placebo
  Arms: Part 3, Arm 2

SUMMARY:
This is a 3-part Phase 2 randomized study evaluating the safety and efficacy of the mutant-selective PI3Kα inhibitor, RLY-2608, in adults and children with PIK3CA Related Overgrowth Spectrum (PROS) and malformations driven by PIK3CA mutation. Part 1 is a dose selection, Part 2 is a basket design with exploratory single-arm cohorts for various subpopulations of participants, and Part 3 is randomized, double-blinded study vs placebo.

ELIGIBILITY:
Key Inclusion Criteria:

* The participant must have a clinical diagnosis of PROS or a malformation within the ISSVA classification.
* One or more documented activating PIK3CA mutation(s) that are targeted by selective PI3Kα inhibitors in lesional tissue and/or cell-free DNA from the lesion or blood. Some participants may be eligible without a documented PIK3CA mutation as long as no other genetic driver has been documented.
* Lansky (<16 yo) or Karnofsky (≥16 yo) performance status of ≥50.
* Agree to provide archived lesional fluid and/or tissue or be willing to undergo pretreatment lesional biopsy (if considered safe and medically feasible) to assess PIK3CA status.

Key Exclusion Criteria:

* History of hypersensitivity to PI3K inhibitors.
* Any factors that increase the risk of QTc prolongation or risk of arrhythmic events
* Clinically significant, uncontrolled cardiovascular disease
* Received disease-directed therapy prior to the first dose of study drug:

  1. Systemic therapy or antibody within 5 half-lives of the therapy.
  2. Local therapy including radiation, surgery, or other procedures within 28 days; lesion(s) must have demonstrated progression after the procedure.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 277 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2031-07 (Estimated); Study Completion 2031-10 (Estimated)

PRIMARY OUTCOMES:
Parts 1 and 2: Determination of a recommended phase 2 dose RP2D(s) for Groups 1, 2, and 3 | Cycle 1 of treatment and at the end of every cycle until study discontinuation
Parts 1 and 2: Occurrence/frequency of Adverse Events (AEs), changes in vital signs, ECGs, and safety laboratory tests and their relationship to the study drugs (safety and tolerability). | Cycle 1 of treatment and at the end of every cycle until study discontinuation
Part 3: Percentage of participants with volumetric Response. | Baseline, Week 24

SECONDARY OUTCOMES:
Part 1 and 2: Percent change from baseline in lesion volume | Baseline, Week 24
Part 1 and 2: Duration of response, defined as the time of first documented response to the date of first documented disease progression or death due to any cause | Approximately every 3 months for approximately the first year, and then every 6 months during treatment
Part 1 and 2: Percentage of participants with volumetric response | Baseline, week 12, week 24
Part 1 and 2: Plasma concentrations and PK parameters of RLY-2608 | Approximately every 2 weeks in Cycle 1, then again at Cycles 2, 4 and Cycle 7 depending on the participant's group
Part 1 and 2: PIK3CA mutational status in lesional fluid and/or tissue | Prior to enrollment
Part 3: Percentage of participants with improvement compared to baseline based on PGI-S, PGI-C and IGIC | Approximately once a month until end of treatment
Part 3: Change from baseline by age-appropriate PROMIS Profile | Approximately once a month until end of treatment
Part 3: Change from baseline in EQ-5D, EQ-5D-Y, or EQ-5D-Y Proxy | Approximately once a month until end of treatment
Part 3: Percent change from baseline in lesion volume | Approximately every 3 months for approximately the first year, and then every 6 months during treatment

CONTACTS AND LOCATIONS:
Locations (25):
- United States (17):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of California, Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of California, San Francisco, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's Hospital of Atlanta, Atlanta, Georgia
  - Riley Children's Hospital, Indianapolis, Indiana
  - Johns Hopkins Medical Institute, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Children's, Cleveland, Ohio
  - Texas Children's Hospital, Houston, Texas
  - University of Wisconsin, Madison, Madison, Wisconsin
- Australia (3):
  - Sydney Children's Hospital, Randwick, Randwick, New South Wales
  - Monash Health, Clayton, Victoria
  - Murdoch Children's Research Institute, Parkville, Victoria
- UC Louvain, Ottignies-Louvain-la-Neuve, Belgium
- Ospedale Pediatrico Bambino Gesù IRCCS, Roma, Italy
- Spain (2):
  - Hospital Sant Joan de Deu, Barcelona
  - Hospital Universitario La Paz, Madrid
- Great Ormond Street Hospital for Children, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No